CLINICAL TRIAL: NCT03850821
Title: Social Mechanisms for Promoting Physical Activity in After School Programs for Underserved Middle School Youth: A Feasibility Trial
Brief Title: Social Mechanisms for Promoting Physical Activity in After School Programs for Underserved Middle School Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nicole Zarrett, Associate Professor of Psychology, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00037559; R21HD077357 (NIH)
Record Dates: First submitted 2018-12-05; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Physical Activity; Obesity Prevention
Keywords: Physical Activity; Community-based Intervention; Social Motivational Theories; Behavioral Change; Social Mechanisms
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized study design will be implemented in which 6 ASPs are randomly assigned to either the Connect Social Mechanisms intervention condition or the active-wait list control condition (8-week intervention, with a 2 week post-intervention data collection).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect Social Mechanisms Intervention (Experimental): The primary components of the intervention included: "Get-to-know-you" sessions aimed specifically at providing youth guided social opportunities to foster friendships, group belonging, and social skills, and novel socially-oriented 'PA sessions' infused within the daily time slot that ASPs' allocated towards recreation. Drawing from theoretical models of motivation, and the investigators' previous ASP studies, key essential elements were identified for facilitating improvements in targeted PA social mechanisms (i.e., friendships, group belonging, and staff connection) and included: 1) social-emotional goal-oriented support, 2) collaborative/cooperative play centered on friendship and informal fun; 3) equal treatment/access, and; 4) inclusive and engaging.
  Interventions: Behavioral: Connect Social Mechanisms Intervention
- Typical ASP curriculum wait-list control (No Intervention): No intervention was implemented within the active wait-list control condition, which served as the typical ASP curriculum control/comparison. After completion of the 8-week intervention (12 weeks including baseline and post-intervention data collection), the control condition received the social mechanisms curriculum as a token of appreciation for participating in measurement.

INTERVENTIONS:
Behavioral: Connect Social Mechanisms Intervention — The "Get-to-Know-You" small group sessions (30 minutes) were designed to increase friendship building skills and involved interactive student-led discussions and activities designed to foster the assets needed to build and support friendships, group cohesion, and staff connections through PA. The PA component of the program (60 minutes) was designed to promote a positive PA social experience and meet youth social affiliation goals. Available games to choose from were novel, inclusive, emphasized teamwork, and centered on social goals. Three different PA stations were offered each program day in which youth rotated. One day each week was designated as a "choice day", whereby youth activity preference ratings were used to determine which activities were offered that day.
  Arms: Connect Social Mechanisms Intervention

SUMMARY:
The primary goal of the Connect feasibility trial was to develop and test the feasibility of a physical activity (PA) social-climate-based intervention within pre-existing after school programs (ASPs) that targets youth social goals (e.g., building friendships through PA) and social competencies (e.g., friendship-building skills) to increase the positive PA affect, cognitions, and moderate-to-vigorous (MV) PA of underserved (i.e., low income, minority status) middle school youth. The 8-week intervention was designed to improve several key social mechanisms within ASPs overlooked in previous interventions (e.g., developing friendship and connection to peers and staff through PA; group belonging, including positive peer PA norms and tangible support) that are key predictors of youth PA and included: 1) "Get to know you" sessions aimed at providing youth guided social opportunities to foster friendship-building skills, and to promote acceptance, cooperation, contribution, and friendship affiliation, and; 2) a novel socially-oriented physical activity curriculum tailored to meet the social goals and needs of program staff and participating youth. Comparison of ASPs receiving the 8-week "Connect" intervention (N=3 ASPs) with ASPs randomized to receive the general ASP curriculum (wait-list control condition; N=3 ASPs) will yield preliminary data on the effectiveness of social mediators for improving moderate-to-vigorous physical activity (MVPA) and preventing obesity among at-risk youth that can inform future intervention design and youth programming policy. Results of this proposed project will provide the basis for conducting a large scale efficacy trial.

First, it is hypothesized that the Connect program will be documented to be feasible as shown by: 1) youth's greater perceived connectedness and PA affiliation goal orientation from baseline to post-intervention; 2). changes in targeted social climate components from baseline to post-intervention as measured by systematic observations, and; 3) adequate dose and fidelity of program implementation as indicated by weekly process evaluations. Second, it is hypothesized that youth in the social climate program (vs. comparison) demonstrate greater increases in positive PA affect, cognitions, and MVPA from baseline to post-intervention.

DETAILED DESCRIPTION:
Physical inactivity has been identified as a primary contributor of childhood obesity and related diseases, with underserved youth (minority and low-income status) at greatest risk of inactivity and its health consequences. However, physical activity (PA) interventions have attained limited-to-no sustained behavior change and thus, have rarely affected targeted physiological or anthropometric health outcomes. Extensive research on participation motivation in sport and physical education shows highly engaged youth report an affiliation orientation towards PA, identifying social reasons and goals (e.g., being with, and making friends) as their primary motivations for participation, and defining PA competence as achieving these social goals. Despite substantial research noting the importance of social goals on PA-based self-determined motivation and participation, PA-based interventions have almost exclusively emphasized approaches centered on constructs related to physical ability (e.g., mastery, self-efficacy). To date, little research has focused on understanding the contributions that affiliation orientations (social goals) make toward promoting sustained youth PA. The investigators argue that adolescents' desire for social connections is a primary goal of action underpinning their PA behavior and thus, a key mechanism to target for sustained behavior change. The Active by Choice Today (ACT) program, conducted by the investigative team is one of the first after school programs (ASPs) to implement a climate-based intervention based on Self-Determination theory that showed significant improvements in PA in underserved youth. However, limited sustained effects found post-intervention, and data from interviews with ACT staff and youth which indicated the presence of several interpersonal barriers (e.g., cliques, teasing) to program effectiveness, suggests additional socially-based climate components still need to be addressed. Systematic observations of ASPs using an observational tool that the PI has developed and tested and additional interviews conducted with ASP staff and youth further suggests that targeting youth social goals (e.g., building friendships through PA) and social competencies (e.g., Friendship-building skills) may be particularly effective for increasing and sustaining the PA of underserved youth. Thus, the proposed study aims to test the feasibility of augmenting the Active by Choice Today (ACT) program through the addition of three key "PA affiliation orientation" elements shown by previous research to be particularly important to adolescents within physical domains: 1) Connecting strengthened friendships to increased PA (developing youth social skills and providing a PA environment that emphasizes friendship building as the goal of PA), 2) Improving peer connectedness and group belonging through PA participation, and 3) Improving interpersonal connections with ASP staff through PA participation. These elements have not been explored in prior research. Enhancing ACT to include these elements in the resultant ACT version 2-Connect intervention is expected to lead to sustained positive PA affect, cognitions, and behaviors in underserved youth. Comparison of ASPs receiving the "Connect" intervention (N=3 ASPs) with ASPs randomized to receive the general ASP curriculum (control condition; N=3 ASPs) will yield preliminary data on the effectiveness of social mediators for improving moderate-to-vigorous (MV)PA and preventing obesity among at-risk youth that can inform future intervention design and youth programming policy. Results of this proposed project will provide the basis for conducting a large scale efficacy trial.

Specific Objectives:

Apply essential social climate elements identified from interviews and the investigators' previous research to design and test the feasibility of the 8-week "Connect" social climate intervention for increasing PA affect, cognition, and MVPA of underserved youth within ASPs.

Primary Aims (Program Development and Feasibility):

1. Through qualitative interviews with program staff and youth at 4 ASP sites serving at-risk youth: a) identify conceptual constructs most relevant for facilitating and supporting youth PA social affiliation goals; b) determine the barriers present within ASPs for meeting youth PA social goals, and; c) obtain staff/youth input on the feasibility and acceptability of initially- developed program components.
2. Explore the feasibility of the Connect program. The Connect program will be documented to be feasible in these ASP programs as shown by: 1) youth's greater perceived connectedness and affiliation goal orientation toward PA from baseline to 12- weeks post-intervention; 2). changes in targeted social climate components from baseline to post-intervention as measured by systematic observations, and; 3) adequate dose and fidelity of program implementation as indicated by weekly process evaluations.

Secondary Aims (Document the preliminary impact of the Connect program on PA outcomes):

1. Assess whether youth in the social climate program (vs. comparison) demonstrate greater increases in positive PA affect, cognitions, and MVPA from baseline to 2-weeks post-intervention.
2. Explore whether youth in the social climate program (vs. comparison) demonstrate healthier BMI trajectories (e.g., slight reduction) from baseline to 2-weeks post-intervention.
3. Assess whether changes in targeted social mechanisms will mediate the effects of the intervention on changes in PA affect, cognitions, and MVPA from baseline to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be currently enrolled in the after school program
* Have parental consent to participate
* Agree to study participation (assent)
* Be available for baseline and post-intervention measurement

Exclusion Criteria:

* Have a medical condition that would interfere with the prescribed physical activity intervention plan
* Have a developmental delay or are in treatment for a psychiatric disorder such that the intervention materials/measures will not be appropriate

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Greater increases (change) in MVPA (using 7-day omni-directional accelerometers) of youth receiving the Connect Social Mechanisms intervention compared to the typical ASP curriculum control. | Baseline to 8 week endpoint
  Objective assessments of PA will be obtained on youth with omni- directional accelerometers. Data will be recorded in 30-s epochs to best capture short bouts of vigorous activity and raw activity data will be converted into time spent in light PA (1.6-2.9 metabolic equivalents (METS); count cut points=100 and 1500 for youth) and moderate-to-vigorous (MV)PA (3-8.9 METS; counts ≥ 1500 for youth) based on activity count thresholds for youth identified by Puyau and colleagues. Youth and staff will wear the belts for one full week at baseline, and again at the 8 wk intervention endpoint.

SECONDARY OUTCOMES:
Greater improvements (change) in the Social Mechanisms intervention ASPs compared to control ASPs in targeted social mechanisms within the ASP for promoting physical activity using a social climate observation tool. | Baseline to 8 week endpoint
  Systematic observations will be conducted using the System for Observing Children's Activity and Relationships during Play (SOCARP) which includes a social climate supplement (MCOT-PA) developed by the PI. Key social mechanisms observed include youth peer interactions and social behaviors (e.g., prosocial interactions like praising peers, antisocial interactions like teasing/bullying), staff behaviors and interactions with youth (e.g., providing praise; engaging in PA with youth), and the nature of program activities for supporting connection and belongingness (e.g., inclusive). Consistent with other PA interventions, teams of two coders will make continuous observations of daily activities throughout 5 days at each ASP at baseline, 4wk midpoint, 8wk endpoint.
Greater improvements (change) in targeted youth PA-based social motivational outcomes of youth receiving the Connect Social Mechanisms intervention compared to the Typical ASP control. | Baseline to 2 weeks post-intervention
  Changes in social, cognitive, and affective components of youth PA motivations will be assessed. Improvements in PA social motivations will be measured using The Social Motivational Orientations Scale for Sport (SMOSS) which assesses youth's social affiliation orientation toward PA (7 items; 5pt scale: 1=strongly disagree, 5=strongly agree; M=2.44; SD=1.04; reliability coefficients range from .77 to .87), with higher mean scores on the affiliation sub scale indicating greater affiliation goals for PA participation.
Greater improvements (change) in targeted youth PA-based cognitive motivational outcomes of youth receiving the Connect Staff-based PA intervention compared to the Typical ASP curriculum control. | Baseline to 2 weeks post-intervention
  Changes in social, cognitive, and affective components of youth PA motivations will be assessed. Youth cognitive components of PA motivation will be assessed using the Treatment Self-Regulation Questionnaire (15 items; 7pt scale: 1=not at all true for me [not autonomously regulated], 7=very true for me; reliability coefficient= .73) autonomous motivation/regulation for exercise, with higher mean scores across scale items indicating greater autonomous regulation.
Greater improvements (change) in targeted youth PA-based social motivational outcomes of youth receiving the Connect Social Mechanisms intervention compared to the Typical ASP curriculum control. | Baseline to 2 weeks post-intervention
  Changes in social, cognitive, and affective components of youth PA motivations will be assessed. The Affective component of motivation will be assessed using The Intrinsic Interest and Regulatory Motives Scale (reliability coefficients from .83 to .94; 5-pt scale: 1=very false [does not enjoy], 5= very true; M=3.7, SD=1.0) with higher mean scores across scale items indicating youth greater intrinsic enjoyment and degree of affective engagement in exercise.
Greater improvements (change) in youth-staff PA-based social connections for promoting physical activity among youth receiving the Connect Social Mechanisms intervention compared to the Typical ASP curriculum control. | Baseline to 2 weeks post-intervention
  Changes in youth PA-based social connections will be measured at three levels: youth-staff connections, peer social connections, and peer support for PA. The Perceived teacher support scale (reliability coefficient =.84; 5-pt scale: 1=completely false [not supportive relationship], 5=completely true [very supportive relationship]; M=3.22; SD=1.05) will be used to evaluate improvements in staff-youth connections, with higher mean scores across the scale items indicating higher quality staff-youth connections.
Greater improvements (change) in youth PA-based peer social support among youth receiving the Connect Social Mechanisms intervention compared to youth in the Typical ASP curriculum control. | Baseline to 2 weeks post-intervention
  The Social Support and Exercise Survey (reliability coefficients= .80-.87; short form, 4 items; 5pt scale: 1=never [receive support], 5=very often [receive support]) will be used to measure increases in youth PA-based peer social support, with higher mean scores indicating greater peer support for PA.
Greater improvements (change) in youth PA-based positive peer connections among youth receiving the Connect Social Mechanisms intervention compared to youth in the Typical ASP curriculum control. | Baseline to 2 weeks post-intervention
  The Peer Motivational Climate in Youth Sport Questionnaire (reliability coefficients=.69-.82; 5-pt scale: 1-completely false, 5=completely true; M=3.18, SD=1.32) will be used to measure youth perceptions peer connections within the program, with higher mean scores across scale items indicating greater positive peer connections.
4. Document the feasibility of the Connect program through adequate dose and fidelity of program implementation as indicated by weekly process evaluation. | week 1 to week 8 of the intervention
  A process evaluation observational tool developed and tested by the PI that monitors dose and fidelity will be conducted within both the intervention and control conditions once a week by an independent process evaluator for the duration of the program. Through observation and use of a quantitative checklist and rating system, the process evaluator will assess whether there are any changes in the structure, delivery, or climate of the control condition, and whether the social climate of intervention ASPs achieve the program's essential elements.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Zarrett, PhD, Principal Investigator — University of South Carolina

REFERENCES:
- [Derived] Zarrett N, Wilson DK, Sweeney A, Bell B, Fairchild AJ, Pinto BM, Miller C, Thames T. An overview of the Connect through PLAY trial to increase physical activity in underserved adolescents. Contemp Clin Trials. 2022 Mar;114:106677. doi: 10.1016/j.cct.2022.106677. Epub 2022 Jan 17. PMID 35051662
- [Derived] Zarrett N, Law LH, Wilson DK, Abraczinskas M, Taylor S, Cook BS, Roberts A. Connect through PLAY: a randomized-controlled trial in afterschool programs to increase adolescents' physical activity. J Behav Med. 2021 Jun;44(3):379-391. doi: 10.1007/s10865-021-00206-0. Epub 2021 Mar 7. PMID 33677766

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03850821/Prot_SAP_000.pdf